CLINICAL TRIAL: NCT03932253
Title: A Single-arm Phase Ia/Ib Study to Evaluate the Safety, Tolerability, PK Characteristics and Anti-tumor Activity of FCN-159 in Patients With Advanced Melanoma Harboring NRAS Aberration(Ia)and NRAS/NF1 Mutation(Ib)
Brief Title: MEK Inhibitor FCN-159 To Treat Advanced Melanoma With NRAS-aberrant (Ia) and NRAS-mutant (Ib)or NF1-mutant(1b)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor R&D strategy adjustment
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-159-001
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1a：0.2 mg, 0.5 mg, 1 mg, 2 mg, 4 mg, 6 mg，8mg, 12mg, 15mg.1b(NRAS),1b(NF1) (Experimental): 1a dose-escalation phase: 9 dose groups during the dose-escalation phase, 0.2 mg, 0.5 mg, 1 mg, 2 mg, 4 mg, 6 mg,8mg, 12mg and 15mg orally, continuous once a day for 28 days a cycle. 1b dose-extension phase: 12mg orally,continuous once a day for 28 days a cycle.
  Interventions: Other: FCN-159

INTERVENTIONS:
Other: FCN-159 — Administered orally once a day

SUMMARY:
Melanoma is one of the most common cutaneous cancers worldwide. Activating mutations in RAS oncogenes are found in a third of all human cancers and NRAS mutations are found in 15%-20% of melanomas. Acquisition of a functional mutation in NRAS results in activation of the Ras / Raf / MEK / ERK signaling pathway leading to unconstrained cell growth and cell transformation. NRAS mutation status was identified as an independent poor prognostic factor in stage IV melanoma. No drug was approved to treat melanoma patients with NRAS mutation or amplification until now. FCN-159, an oral and potent MEK1/2 inhibitor, has more than 10 folds higher selectivity against activated MEK1 and MEK2 compared with trametinib, and has demonstrated significant antitumor growth inhibition in two patient-derived xenograft (PDX) models with NRAS mutation. Approximately 10%-15% of melanomas is reported to be NF1-mutant. NF1 gene is located in chromosome 17 q11.2 and encodes neurofibromin 1. Neurofibromin 1 is a RAS-specific GTP enzyme-activated protein that converts RAS from the active guanosine triphosphate (GTP) binding state to the inactivated guanosine diphosphate (GDP) binding state and acts as a negative regulatory factor for RAS and its downstream MAPK and PI3K-Akt pathways. Recent treatments of NF1 mutation focus on the downstream of the MAPK pathway, such as MEK kinase. Blocking the MEK kinase can reduce neurofibroma in mice with NF1 mutation and prolong the survival time of mice with malignant peripheral nerve sheath tumor (MPNST) xenograft. In the NF1 mutant monocytic leukemia mouse model, the use of MEK inhibitors can improve mouse survival rate. This is the first in human study to evaluate the safety and anti-tumor activity in patients.

DETAILED DESCRIPTION:
This is a phase Ia/Ib, open label, dose-escalation and dose-expansion study that will evaluate the safety, pharmacokinetics (PK), and preliminary anti-tumor activity of FCN-159 in up to 85 patients with NRAS-aberrant including both NRAS amplification and mutation (Ia) and NRAS-mutation (Ib) or NF-1 mutation (Ib) in local advanced or metastatic melanoma. In this study, the dose escalation phase utilizes accelerated titration design (switch to 3+3 mode once a grade≥2 AE is reported) with starting dose of 0.2 mg, QD, orally, and the dose will be escalated up to Maximum-Tolerated Dose (MTD) or until the Recommended Phase 2 dose (RP2D) is identified. The dose level will be considered to expand up to 6 patients if the objective response is observed, intends to collect more clinical data to support the RP2D determination. After the MTD or RP2D dose is identified, dose expansion stage (Phase Ib) is conducted to further evaluate the safety and efficacy of FCN-159 in patients with NRAS-mutant (Cohort 1) or NF1-mutant melanoma (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, 18-70 years old (Ia); 18 years old and above (Ia expansion part & phase Ib);
2. Histologically or cytologically diagnosed advanced melanoma who cannot be surgically resected, stage III or IV, and have failed or rejected standard treatment;
3. Written report of NRAS aberrant (Ia) or NRAS mutation (Ib) or NF1 mutation (Ib);
4. ECOG 0 or 1;
5. Expected survival of at least 12 weeks;
6. Adequate organ functions;
7. At least one measurable lesion per RECIST v1.1 criteria.
8. Able to understand and sign consent form.
9. For female patients or partners with fertility: maintain abstinence.

Exclusion Criteria:

1. Radiotherapy, major surgery, mono-clone antibody targeted therapy, immunotherapy or other treatment within 4 weeks prior to enrollment.
2. Chemotherapy and small molecule targeted therapy within 2 weeks of enrollment.
3. Participated in other clinical trials within 4 weeks prior to enrollment or 5 T1/2;
4. Previous usage of MEK inhibitor;
5. Uncontrolled central nervous system metastasis or injury.
6. Unrecovered >grade 2 AE caused by previous anti-tumor therapy;
7. Strong inhibitors/inducers of CYP3A4, CYP2C8 or CYP2C9 within 14 days prior to the start of dosing.
8. Taking drugs that prolong QTc interval;
9. Dysphagia, or active digestive system disease, or malabsorption syndrome, or other conditions affecting FCN-159 absorption.
10. Previous or current retinal vein stenosis, retinal detachment, central retinal vein occlusion, glaucoma.
11. Interstitial pneumonia, including clinically significant radiationpneumonitis.
12. Insufficient cardiac function or disease;
13. Pregnant or lactating woman.
14. Known to be allergic to any excipients of FCN-159.
15. Clinically active infections;
16. Significant active disease that in the investigator's opinion would adversely impact on his/her participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 1 month.
  To assess safety and tolerability of FCN-159 with a maximum tolerated dose (MTD) in patients with advanced melonoma.
Objective response rate（ORR) | through study completion, an average of 1 year.
  The proportion of confirmed complete response (CR) or partial response (PR) patients evaluated according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. in patients with unresectable stage III or IV melanoma with NRAS mutation or NF1 mutation.

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs) | through study completion, an average of 1 year.
  All subjects , assessment according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0.
PFS in months | through study completion, an average of 1 year.
  To assess the efficacy of FCN-159 monotherapy in patients with unresectable stage III or IV melanoma with NRAS mutation or NF1 mutation.
OS in months | through study completion, an average of 1 year.
  To assess the efficacy of FCN-159 monotherapy in patients with unresectable stage III or IV melanoma with NRAS mutation or NF1 mutation.
1-year OS rate(%) | through study completion, an average of 1 year.
  To assess the efficacy of FCN-159 monotherapy in patients with unresectable stage III or IV melanoma with NRAS mutation or NF1 mutation.
DoR in months | through study completion, an average of 1 year.
  To assess the efficacy of FCN-159 monotherapy in patients with unresectable stage III or IV melanoma with NRAS mutation or NF1 mutation.
CBR in months | through study completion, an average of 1 year.
  To assess the efficacy of FCN-159 monotherapy in patients with unresectable stage III or IV melanoma with NRAS mutation or NF1 mutation.
AUC(0-last) | 1 month.
  Pharmacokinetics of FCN-159
AUC(0-∞) | 1 month.
  Pharmacokinetics of FCN-159
Cmax | 1 month.
  Pharmacokinetics of FCN-159
Tmax | 1 month.
  Pharmacokinetics of FCN-159
t1/2 | 1 month.
  Pharmacokinetics of FCN-159
CL/F | 1 month.
  Pharmacokinetics of FCN-159
RAUC | 1 month.
  Pharmacokinetics of FCN-159
RCmax | 1 month.
  Pharmacokinetics of FCN-159

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mao L, Guo J, Zhu L, Jiang Y, Yan W, Zhang J, Hui AM, Yang Y, Diao L, Tan Y, Zhao H, Jiang Y, Wu Z, Si L. A first-in-human, phase 1a dose-escalation study of the selective MEK1/2 inhibitor FCN-159 in patients with advanced NRAS-mutant melanoma. Eur J Cancer. 2022 Nov;175:125-135. doi: 10.1016/j.ejca.2022.08.005. Epub 2022 Sep 13. PMID 36113242